CLINICAL TRIAL: NCT03980275
Title: Selective Laryngeal Reinnervation for Bilateral Vocal Fold Paralysis
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 1806019347
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Bilateral Vocal Cord Paralysis
Keywords: Bilateral vocal fold paralysis; Tracheostomy dependency; Glottic airway obstruction; Stridor
MeSH Terms: conditions — Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study examining the treatment outcomes of selective laryngeal reinnervation procedures for patients with bilateral vocal fold paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70
* Patients with bilateral vocal fold paralysis without any improvement for 6 months

Exclusion Criteria:

* Patients with neck or chest radiation
* Patients with severe respiratory compromise
* Patients with cricoarytenoid ankylosis
* Patients with pacemakers
* Patients who are pregnant
* Patients with cochlear implant, or any nerve stimulator implants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with bilateral vocal fold paralysis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in breathing function is being assessed and measured by the Dyspnea Index (DI) | Pre-surgery and then post-surgery at 1 week, 1 month, 3 months and every 3 months thereafter up to 18 months, then at 24 months
  The DI is a standardized and validated tool to quantify patients' symptoms of upper airway dyspnea. It's a 10-item questionnaire. The lowest score is 0, which indicates that the patient is never experiencing dyspnea symptoms, and the highest is 40, which indicates that the patient is always experiencing dyspnea symptoms.
Change in breathing function is being assessed and measured by pulmonary function testing | Pre-surgery and then post-surgery at 1 week, 1 month, 3 months and every 3 months thereafter up to 18 months, then at 24 months
  Pulmonary function testing will measure the total inspiratory and expiratory tidal volumes.

CONTACTS AND LOCATIONS:
Overall Officials: Babak Sadoughi, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Sean Parker Institute for the Voice, New York, New York, United States